CLINICAL TRIAL: NCT04309656
Title: An Open-label, Randomized, Four-period, Crossover Study in Two Panels of Healthy Adult Subjects to Assess the Relative Bioavailability, Food Effect, and Dose-dependence of Single-dose Immediate-release and Single-dose Dispersible Formulations of Pretomanid
Brief Title: Single-dose Study in Two Panels of Healthy Adult Participants to Assess Immediate-Release and Dispersible Formulations of Pretomanid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pa-824-CL-011
Record Dates: First submitted 2020-01-23; First posted 2020-03-16 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Multi-drug Resistant Tuberculosis
Keywords: MDR-TB (multi-drug resistant tuberculosis); Extensively Resistant Pulmonary Tuberculosis; XDR-TB (extensively drug resistant tuberculosis); pretomanid; PA-824
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis | interventions — pretomanid

STUDY DESIGN:
Intervention Model Description: Each panel of 24 subjects will be randomized according to the same 4-sequence, 4-period Williams design, in which each participant will receive four single-dose treatments. Subjects in Panel 1 will receive all treatments after consuming an FDA standard high-fat, high-calorie breakfast following an overnight fast of at least 10 hours. Subjects in Panel 2 will receive all treatments directly following an overnight fast of at least 10 hours. The two panels will be investigated concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panel 1: Pretomanid after meal (Experimental): Each participant will receive four single-dose treatments with a 7-day washout period between each dose. Panel 1 will receive a meal before dosing.
  Interventions: Drug: Pretomanid
- Panel 2: Pretomanid after fast (Experimental): Each participant will receive four single-dose treatments with a 7-day washout period between each dose. Panel 2 will fast before dosing.
  Interventions: Drug: Pretomanid

INTERVENTIONS:
Drug: Pretomanid — 1. Treatment A (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
  2. Treatment B (test) = 200 mg given as four 50-mg tablets (using the dispersible pediatric formulation), orally administered.
  3. Treatment C (test) = single 50-mg dispersible tablet, orally administered.
  4. Treatment D (test) = single 10-mg dispersible tablet, orally administered.
  Other Names: PA-824

SUMMARY:
This is a single-dose, open-label, randomized, four-period, four-treatment, crossover study in healthy adult subjects.

DETAILED DESCRIPTION:
This is a single-dose, open-label, randomized, four-period, four-treatment, crossover study in healthy adult subjects. Each panel of 24 subjects will be randomized according to the same 4-sequence, 4- period Williams design, in which each participant will receive four single-dose treatments. Subjects in Panel 1 will receive all treatments after consuming an FDA standard high-fat, high-calorie breakfast following an overnight fast of at least 10 hours. Subjects in Panel 2 will receive all treatments directly following an overnight fast of at least 10 hours. The two panels will be investigated concurrently.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female. Females must not be pregnant or breastfeeding.
* Willing and able to comply with the contraception requirements.
* Between 19 and 50 years of age (inclusive) at the time of screening.
* Body mass index (BMI) between 18.50 and 32 kg/m2 (inclusive) and weighs a minimum of 50 kg.

Key Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* Vital signs at screening (measured sitting after a minimum 3 minutes rest) as follows: blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg or a heart rate lower than 40 bpm or higher than 99 bpm. Out-of-range vital signs may be repeated once.
* History or presence of allergic or adverse response to pretomanid or related drugs.
* Use of any drugs or treatment with any known drugs that are moderate or strong inducers or inhibitors of cytochrome P450 (CYP) enzymes (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine) and/or P-gp, including St. John's Wort, within 30 days before the first dose of study medication, and that, in the Investigator's judgment, may impact subject safety or the validity of the study results.
* Female with a positive pregnancy test result.
* Positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.
* Hemoglobin <10.0 g/dL.
* ALT (alanine transaminase) or AST (aspartate aminotransferase) >2.0 x the upper limit of normal (ULN).
* Hyperbilirubinemia >1.5 x ULN.
* History or presence of alcoholism or drug abuse within the past 2 years as determined by the Investigator to be clinically relevant.
* Any clinically significant electrocardiogram abnormality at Screening (as deemed by decision of the Investigator and the Study Sponsor's Medical Monitor).
* QTcF interval >450 msec for males or >470 msec for females at screening, Day -1, or Day 1 (pre-dose), or history of prolonged QT syndrome.
* Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease, congestive heart failure or terminal cancer).

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lombardi, MD, Study Director — TB Alliance
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States

REFERENCES:
- [Derived] Zou Y, Nedelman J, Lombardi A, Pappas F, Karlsson MO, Svensson EM. Characterizing Absorption Properties of Dispersible Pretomanid Tablets Using Population Pharmacokinetic Modelling. Clin Pharmacokinet. 2022 Nov;61(11):1585-1593. doi: 10.1007/s40262-022-01163-w. Epub 2022 Sep 30. PMID 36180816

RESULTS

PARTICIPANT FLOW:
Groups:
- Panel 1: Pretomanid After Meal: Each participant will receive four single-dose treatments. Panel 1 will receive a required FDA standard high fat, high-calorie meal before dosing.
  Pretomanid: 1) Treatment A (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
  2) Treatment B (test) = 200 mg given as four 50-mg tablets (using the dispersible pediatric formulation), orally administered.
  3) Treatment C (test) = single 50-mg dispersible tablet, orally administered. 4) Treatment D (test) = single 10-mg dispersible tablet, orally administered.
- Panel 2: Pretomanid After Fast: Each participant will receive four single-dose treatments. Panel 2 will fast before dosing.
  Pretomanid: 1) Treatment A (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
  2) Treatment B (test) = 200 mg given as four 50-mg tablets (using the dispersible pediatric formulation), orally administered.
  3) Treatment C (test) = single 50-mg dispersible tablet, orally administered. 4) Treatment D (test) = single 10-mg dispersible tablet, orally administered.
Period: Overall Study
Arm/Group | Panel 1: Pretomanid After Meal | Panel 2: Pretomanid After Fast
Started | 24 (All 24 participants received Treatments A, B, C and D) | 24 (All 24 participants received Treatments A, B, C and D)
Completed | 24 (All 24 participants received Treatments A, B, C and D) | 24 (All 24 participants received Treatments A, B, C and D)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panel 1: Pretomanid After Meal: Each participant will receive four single-dose treatments. Panel 1 will receive a required FDA standard high fat, high-calorie meal before dosing.
- Panel 2: Pretomanid After Fast: Each participant will receive four single-dose treatments. Panel 2 will fast before dosing.
- Total: Total of all reporting groups
Arm/Group | Panel 1: Pretomanid After Meal | Panel 2: Pretomanid After Fast | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (8.5) | 36.4 (7.2) | 37.0 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 11 | 16 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 15 | 23
  White | 14 | 9 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Height at Screening [Mean (Standard Deviation); unit: centimeter] | 170.70 (7.962) | 170.96 (11.953) | 170.83 (10.048)
Weight at Screening [Mean (Standard Deviation); unit: kilogram] | 79.06 (11.601) | 78.49 (13.633) | 78.77 (12.526)
BMI at Screening [Mean (Standard Deviation); unit: kilogram per meter squared] | 27.08 (2.882) | 26.76 (2.996) | 26.92 (2.913)

OUTCOME MEASURES:

1. Primary Outcome: Relative Bioavailability - Cmax
Description: Relative bioavailability will be determined separately for each panel using Cmax
Time Frame: intake (pre-dose), and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose
Population: Quantifiable predose concentrations that were below 5% of the respective Cmax values were included in the pharmacokinetic analyses without adjustment. Data for subjects with quantifiable predose concentrations that were above 5% of the respective Cmax values were excluded from concentration-time descriptive statistics and mean concentration-time profiles
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Panel 1: Pretomanid After Meal: Each participant will receive four single-dose treatments. Panel 1 will receive a meal before dosing.
  Pretomanid: 1) Treatment A (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
  2) Treatment B (test) = 200 mg given as four 50-mg tablets (using the dispersible pediatric formulation), orally administered.
  3) Treatment C (test) = single 50-mg dispersible tablet, orally administered. 4) Treatment D (test) = single 10-mg dispersible tablet, orally administered.
Arm/Group | Panel 1: Pretomanid After Meal | Panel 2: Pretomanid After Fast
Number analyzed (Participants) | 24 | 24
ng/mL
  Treatment A | 2170 (484) | 1180 (401)
  Treatment B | 1850 (354) | 1090 (334)
  Treatment C: number analyzed (Participants) | 23 | 23
  Treatment C | 389 (58.8) | 427 (111)
  Treatment D: number analyzed (Participants) | 16 | 18
  Treatment D | 76.7 (14.2) | 110 (20.2)
Statistical Analysis 1: Comparison: Panel 1: Pretomanid After Meal; Test type: Equivalence — Comparisons performed: Treatment B (test) versus Treatment A (reference). Relative bioavailability of test compared to reference assessed via 90% CI. CI obtained by taking the antilog of the upper and lower limits of CI for the difference of the least squares means on the log scale within the ANOVA framework model; p = 0.0001, ANOVA; Geometric mean ratio (%) = 85.85, 90% CI 2-sided [81.21 to 90.75]
Statistical Analysis 2: Comparison: Panel 2: Pretomanid After Fast; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3001, ANOVA; Geometric mean ratio (%) = 92.99, 90% CI 2-sided [82.65 to 104.62]

2. Primary Outcome: Relative Bioavailability - AUC 0-t
Description: Relative bioavailability will be determined separately for each panel using AUC 0-t (area under the time vs concentration curve from time 0 to time t : h*ng/mL)
Time Frame: intake (pre-dose), and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Panel 1: Pretomanid After Meal | Panel 2: Pretomanid After Fast
Number analyzed (Participants) | 24 | 24
h*ng/mL
  Treatment A | 54900 (10700) | 32900 (7580)
  Treatment B | 55200 (10800) | 30200 (9030)
  Treatment C: number analyzed (Participants) | 23 | 23
  Treatment C | 12300 (2790) | 10900 (3150)
  Treatment D: number analyzed (Participants) | 16 | 18
  Treatment D | 2040 (514) | 2460 (513)
Statistical Analysis 1: Comparison: Panel 1: Pretomanid After Meal; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.6686, ANOVA; Geometric mean ratio (%) = 100.60, 90% CI 2-sided [98.23 to 103.03]
Statistical Analysis 2: Comparison: Panel 2: Pretomanid After Fast; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0745, ANOVA; Geometric mean ratio (%) = 89.70, 90% CI 2-sided [81.20 to 99.10]

3. Primary Outcome: Relative Bioavailability - AUC 0-inf
Description: Relative bioavailability will be determined separately for each panel using AUC 0-inf (area under the time vs concentration curve from time 0 to infinite time)
Time Frame: intake (pre-dose), and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Panel 1: Pretomanid After Meal | Panel 2: Pretomanid After Fast
Number analyzed (Participants) | 24 | 24
h*ng/mL
  Treatment A | 57400 (12300) | 34700 (8330)
  Treatment B | 57900 (12400) | 31900 (10200)
  Treatment C: number analyzed (Participants) | 23 | 23
  Treatment C | 12700 (3210) | 11400 (3440)
  Treatment D: number analyzed (Participants) | 16 | 18
  Treatment D | 2100 (552) | 2530 (551)
Statistical Analysis 1: Comparison: Panel 1: Pretomanid After Meal; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.4683, ANOVA; Geometric mean ratio (%) = 101.03, 90% CI 2-sided [98.65 to 103.47]
Statistical Analysis 2: Comparison: Panel 2: Pretomanid After Fast; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0734, ANOVA; Geometric mean ratio (%) = 89.63, 90% CI 2-sided [81.10 to 99.05]

4. Secondary Outcome: Food Effect - Ratio of Cmax Fed Vs Fasted
Description: Food effect on bioavailability will be determined across panels using Cmax.
  Reported in Ratio(%) of the Geometric Mean (Fed)/Geometric Mean (Fasted) based on Least Squares Mean of log-transformed parameter values (ng/mL)
Time Frame: intake (pre-dose), and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose
Population: Ratio(%) = Geometric Mean (Test)/Geometric Mean (Ref). Quantifiable predose concentrations that were below 5% of the respective Cmax values were included in the pharmacokinetic analyses without adjustment. Data for subjects with quantifiable predose concentrations that were above 5% of the respective Cmax values were excluded from concentration-time descriptive statistics and mean concentration-time profiles
Measure: Number (90% Confidence Interval); unit: Ratio (%)
Groups:
- Treatment A Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions
  Pretomanid: 1) Treatment A (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
- Treatment B Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions
  Treatment B (test) = 200 mg given as four 50-mg tablets (using the dispersible pediatric formulation), orally administered.
- Treatment C Fed and Fasted: Each participant will receive four single-dose treatments. Panel 1 will receive a meal before dosing.
  Treatment C (test) = single 50-mg dispersible tablet, orally administered.
- Treatment D Fed and Fasted: Each participant will receive four single-dose treatments. Panel 1 will receive a meal before dosing.
  Treatment D (test) = single 10-mg dispersible tablet, orally administered.
Arm/Group | Treatment A Fed and Fasted | Treatment B Fed and Fasted | Treatment C Fed and Fasted | Treatment D Fed and Fasted
Number analyzed (Participants) | 48 | 48 | 46 | 34
Ratio (%) | 187.65 [165.90 to 212.25] | 173.24 [153.26 to 195.82] | 93.25 [83.16 to 104.56] | 69.38 [61.96 to 77.68]

5. Secondary Outcome: Food Effect - Ratio of AUC 0-t Fed Vs Fasted
Description: Food effect on bioavailability was assessed across panels based on the 90% confidence intervals (CIs) for estimates of the geometric mean ratios between AUC 0-t of fed versus fasted across panels. An analysis of variance was used for each treatment with panel as the fixed effect.
Time Frame: intake (pre-dose), and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Ratio (%)
Groups:
- Treatment A Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions
  Treatment A (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
- Treatment B Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions
  2) Treatment B (test) = 200 mg given as four 50-mg tablets (using the dispersible pediatric formulation), orally administered.
- Treatment C Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions
  Pretomanid: 1) Treatment C (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
- Treatment D Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions
  Pretomanid: 1) Treatment D(reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
Arm/Group | Treatment A Fed and Fasted | Treatment B Fed and Fasted | Treatment C Fed and Fasted | Treatment D Fed and Fasted
Number analyzed (Participants) | 48 | 48 | 46 | 34
Ratio (%) | 167.96 [151.40 to 186.33] | 188.36 [165.60 to 214.26] | 114.09 [99.70 to 130.55] | 81.74 [71.53 to 93.42]

6. Secondary Outcome: Food Effect - Ratio of AUC 0-inf Fed Vs Fasted
Description: Food effect on bioavailability was assessed across panels based on the 90% confidence intervals (CIs) for estimates of the geometric mean ratios between AUC 0-inf of fed versus fasted across panels. An analysis of variance was used for each treatment with panel as the fixed effect
Time Frame: intake (pre-dose), and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose
Measure: Number (90% Confidence Interval); unit: Ratio (%)
Groups:
- Treatment A Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions.
  Treatment A (reference) = 200 mg pretomanid given as a single 200 mg tablet (using the immediate release formulation), orally administered
- Treatment C Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions Treatment C (test) = single 50-mg dispersible tablet, orally administered.
- Treatment D Fed and Fasted: Each participant will receive four single-dose treatments in both fed and fasted conditions Treatment D (test) = single 10-mg dispersible tablet, orally administered.
Arm/Group | Treatment A Fed and Fasted | Treatment B Fed and Fasted | Treatment C Fed and Fasted | Treatment D Fed and Fasted
Number analyzed (Participants) | 48 | 48 | 46 | 34
Ratio (%) | 166.38 [149.07 to 185.69] | 187.54 [163.44 to 215.20] | 113.58 [98.52 to 130.95] | 81.57 [71.07 to 93.61]

7. Secondary Outcome: Adverse Events - Overall Incidence
Description: All listed adverse events (AEs) are treatment emergent adverse events (TEAE) which are defined as AEs that started or worsened at or after the first administration of IMP up to and including
Time Frame: throughout the study, approximately 33 days
Population: All participants randomized
Measure: Count of Participants; unit: Participants
Groups:
- Panel 1: Treatment A; Panel 1: Treatment B; Panel 1: Treatment C; Panel 1: Treatment D: Each participant received four single-dose treatments. Panel 1 received a meal before dosing.
  Pretomanid: 1) Treatment A (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
  2) Treatment B (test) = 200 mg given as four 50-mg tablets (using the dispersible pediatric formulation), orally administered.
  3) Treatment C (test) = single 50-mg dispersible tablet, orally administered. 4) Treatment D (test) = single 10-mg dispersible tablet, orally administered.
- Panel 2:Treatment A; Panel 2: Treatment B; Panel 2: Treatment C; Panel 2: Treatment D: Each participant received four single-dose treatments. Panel 2 fasted before dosing.
  Pretomanid: 1) Treatment A (reference) = 200 mg given as a single 200 mg tablet (using the immediate release formulation), orally administered.
  2) Treatment B (test) = 200 mg given as four 50-mg tablets (using the dispersible pediatric formulation), orally administered.
  3) Treatment C (test) = single 50-mg dispersible tablet, orally administered. 4) Treatment D (test) = single 10-mg dispersible tablet, orally administered
Arm/Group | Panel 1: Treatment A | Panel 1: Treatment B | Panel 1: Treatment C | Panel 1: Treatment D | Panel 2:Treatment A | Panel 2: Treatment B | Panel 2: Treatment C | Panel 2: Treatment D
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants | 5 | 9 | 2 | 6 | 3 | 3 | 1 | 4

ADVERSE EVENTS:
Time Frame: Day 1 to Day 33
Arm/Group | Panel 1: Treatment A | Panel 1: Treatment B | Panel 1: Treatment C | Panel 1: Treatment D | Panel 2:Treatment A | Panel 2: Treatment B | Panel 2: Treatment C | Panel 2: Treatment D
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 5/24 | 9/24 | 2/24 | 6/24 | 3/24 | 3/24 | 1/24 | 4/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel 1: Treatment A (N=24) | Panel 1: Treatment B (N=24) | Panel 1: Treatment C (N=24) | Panel 1: Treatment D (N=24) | Panel 2:Treatment A (N=24) | Panel 2: Treatment B (N=24) | Panel 2: Treatment C (N=24) | Panel 2: Treatment D (N=24)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 3 (4) | 3 (6) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT04309656/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04309656/SAP_001.pdf